CLINICAL TRIAL: NCT01042795
Title: Phase II Trial of Adjuvant Sutent for Patients With High Risk Urothelial Carcinoma After Neoadjuvant Chemotherapy and Cystectomy
Brief Title: Trial of Adjuvant Sutent for Patients With High Risk Urothelial Carcinoma After Neoadjuvant Chemotherapy and Cystectomy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study closed due to poor accrual
Sponsor: University of Michigan (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Cheryl Lee, Associate Professor of Urology, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00030127
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-05

CONDITIONS: Urothelial Carcinoma; Bladder Cancer
Keywords: sunitinib; bladder neoplasm; adjuvant treatment; disease free survival; cystectomy
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Continuous Daily Dosing of Sunitinib (Experimental)
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — Sunitinib 37.5 mg daily X 16 weeks
  Other Names: Sutent

SUMMARY:
The purpose of this study is to determine whether sutent (sunitinib)is effective in preventing tumor recurrence in patients with high risk bladder cancer who have previously had chemotherapy and cystectomy (bladder removal).

A 4 month supply of the drug is given to patients beginning 2-3 months after bladder removal. The patients are followed up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of bladder carcinoma (>50% urothelial carcinoma)
* Prior treatment with at least one cycle of platin-based neoadjuvant chemotherapy
* Prior treatment with radical cystectomy revealing pT3NxM0 or pTanyN+M0
* ECOG performance status of 0-1 (Appendix 2).
* No evidence of metastases within 4 weeks of registration
* Adequate organ and marrow function obtained within 14 days of registration

Exclusion Criteria:

* Severe or uncontrolled acute or chronic medical or psychiatric condition
* Prior antiangiogenic therapy
* Prior pelvic radiation for bladder cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-09; Primary Completion 2012-04 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Dosing Period - 16 Weeks of Daily Doses
Arm/Group | Continuous Daily Dosing of Sunitinib
Started | 7
Completed | 2
Not Completed | 5
Period: Follow up - 22 Months After Drug Start
Arm/Group | Continuous Daily Dosing of Sunitinib
Started | 2
Completed | 0
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Continuous Daily Dosing of Sunitinib
Number analyzed (Participants) | 7
Age, Customized [Count of Participants; unit: Participants]
  18-85 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival
Description: 2-year disease free survival
Time Frame: 2- year
Measure: Number; unit: months
Arm/Group | Continuous Daily Dosing of Sunitinib
Number analyzed (Participants) | 7
months
  Patient 1 Time to Recurrence | 4.7
  Patient 2 Last Follow up. No Recurrence | 21.1
  Patient 3 Time to Recurrence | 21.2
  Patient 4 Last Follow up. No Recurrence | 17.1
  Patient 5 Last Follow up. No Recurrence | 12.3
  Patient 6 Time to Recurrence | 12.2
  Patient 7 Last Follow up. No Recurrence | 9.4

ADVERSE EVENTS:
Time Frame: 21.5 months - after that point no one was still in the trial
Arm/Group | Continuous Daily Dosing of Sunitinib
Serious Adverse Events (participants affected / at risk) | 3/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Continuous Daily Dosing of Sunitinib (N=7)
pyelonephritis (Infections and infestations) | 1
anemia (Blood and lymphatic system disorders) | 1
mucositis (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Continuous Daily Dosing of Sunitinib (N=7)
neutropenia (Blood and lymphatic system disorders) | 6
diarrhea (Gastrointestinal disorders) | 5
nausea (Gastrointestinal disorders) | 5
fatigue (General disorders) | 3
hypertension (Vascular disorders) | 3
thrombocytopenia (Blood and lymphatic system disorders) | 3
cardiac dysfunction (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes